CLINICAL TRIAL: NCT00666744
Title: A Randomised Controlled Trial of Family Mediated Exercises (FAME) Following Stroke
Acronym: FAME
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: Foundation for Medical Research (Other); Friends of the Royal Hospital Donnybrook (Unknown)
Responsible Party: Dr. Emma Stokes, University of Dublin, Trinity College
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 08/19; Irish Heart Foundation - FAME
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Last update posted 2008-10-29 (Estimated); Status verified 2008-04

CONDITIONS: Weakness; Balance
Keywords: exercise; frequency; duration
MeSH Terms: conditions — Asthenia; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Exercise Intervention - additional lower limb exercises will be completed by the person with stroke with the assistance of his/her family for 35 minutes daily for a period of 8 weeks.
  Interventions: Other: Family Mediated Exercise Therapy
- 2 (No Intervention): Participants in this group will receive routine exercise therapy following stroke

INTERVENTIONS:
Other: Family Mediated Exercise Therapy — 35 minutes of lower limb exercises to be completed by the person with stroke on a daily basis with the assistance of their family for a period of 8 weeks.
  Arms: 1

SUMMARY:
The aim of the study is to evaluate the functional recovery in two groups of primary stroke patients presenting with moderate/severe disability over a six month period through the implementation of a randomised controlled trial. The first group or the experimental group will receive routine therapy and additional lower limb exercise therapy in the form of family assisted exercises. The second group or the control group will receive routine therapy with no additional formal input from their family members. A secondary aim of the project is to evaluate the impact of the FAME programme on the person with stroke and the individual (s) assisting in the delivery of exercises.

DETAILED DESCRIPTION:
Participants with primary stroke eligible for inclusion to the study at 2 weeks post stroke will be randomised into either a 'control' group that will receive routine therapy or an 'experimental' group that will receive routine therapy AND additional 'family mediated exercise therapy.

Training will be provided to the nominated family member (s)/friends of participants in the 'intervention' group on a weekly basis by the research physiotherapist (R1). Family members/friends will be requested to keep an exercise diary on a daily basis to document completion of exercises. The trial will continue for eight weeks with an expectation that at least 1200 additional minutes of FAME therapy will be delivered over this time period. Each FAME session is expected to last 35-40 minutes.

Exercises will include repetitive sit to stand exercises with an emphasis on improving symmetry, weight bearing exercises during standing, bridging, straight leg raises, quadriceps strengthening exercises, active/active assisted range of movement exercises for the lower limb and walking. Outcome will be assessed by a blinded outcome assessor (R2) on entry to the study, at eight weeks (post-intervention) and again three months post-intervention (follow-up)

In addition, a semi-structured interview will be carried out with a random sample of the participants and their family member (s)/friends to gain a more qualitative insight into the impact of the programme on those involved. This interview will be completed by a person unknown to the participant. (R3)

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of first unilateral stroke
* Patients who score between 3.2 and 5.2 on the Orpington Prognostic Scale
* Patients participating in a physiotherapy programme
* Patients willing to give informed written consent
* Patients with family willing to participate in their assigned physiotherapy intervention programme

Exclusion Criteria:

* hemiplegia of a non-vascular origin
* discharged from hospital less than two weeks following stroke
* pre-existing neurological disorder
* any lower limb orthopaedic condition that may limit exercise capacity
* aphasia
* cognitive impairment
* not willing to give written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-03 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Fugl Meyer (FM) Assessment | Baseline, post intervention and 3 month follow-up

SECONDARY OUTCOMES:
Berg Balance Scale (BBS) | Baseline, post intervention and 3 month follow-up
Motor Assessment Scale (MAS) | Baseline, post-intervention and 3 month follow up
Six Minute Walk Test (SMWT) | Baseline, post-intervention and 3 month follow up
Barthel Index (BI) | Baseline, post-intervention and 3 month follow up
Re-integration into Normal Living Index (RNLI) | Baseline, post-intervention and 3 month follow up
Nottingham Extended Activities of Daily Living (EADL) | Baseline, post-intervention and 3 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Emma Stokes, PhD, Principal Investigator — University of Dublin, Trinity College; Tara Cusack, PhD, Principal Investigator — University College Dublin
Locations (2):
- Ireland (2):
  - Beaumont Hospital, Dublin
  - MaterMisercordiae University Hospital, Dublin

REFERENCES:
- [Derived] Galvin R, Cusack T, Stokes E. A randomised controlled trial evaluating family mediated exercise (FAME) therapy following stroke. BMC Neurol. 2008 Jun 20;8:22. doi: 10.1186/1471-2377-8-22. PMID 18570643